CLINICAL TRIAL: NCT02166996
Title: A Prospective Comparison of Suture Removal Time for Simple Surgical Defects of the Head and Neck
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sundsvall Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dnr 2011-56-31M
Record Dates: First submitted 2013-03-31; First posted 2014-06-18 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2012-12

CONDITIONS: Cutaneous Tumors
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Suture removal time 7 days.
  Interventions: Procedure: Suture removal time 7 days
- B (Experimental): Suture removal time 14 days.
  Interventions: Procedure: Suture removal time14 days

INTERVENTIONS:
Procedure: Suture removal time 7 days — To compare cosmetic outcome of surgical defects of head and neck, repaired with non-resorbable monofilament nylon sutures from the aspect of suture removal time 7 days.
  Arms: A
Procedure: Suture removal time14 days — To compare cosmetic outcome of surgical defects of head and neck, repaired with non-resorbable monofilament nylon sutures from the aspect of suture removal time 14 days
  Arms: B

SUMMARY:
A single-center, prospective, randomized comparison with blinded assessment of cosmetic outcome.

To compare cosmetic outcome of surgical defects of head and neck, repaired with non-resorbable monofilament sutures from the aspect of suture removal time 7 and 14 days. Data are gathered through a standardized form at the time of surgery concerning width and length of the surgical excisions, and if the patient has any systemic cortisone treatment or diabetes mellitus. At the time of surgery the patients are randomised to a suture time at 7 or 14 days postoperatively and all receive the same written information about postoperative care and restrictions.

Photographs of the scars are taken one month and one year after the procedure and rated using a visual analogue scale (VAS) by three independent assessors blinded to the intervention and suture time. The width of the scar is measured after one ear.

Study hypothesis is that leaving non-resorbable monofilament sutures in clean surgical wounds in the head and neck area for up to 14 days does not lead to poor cosmetic outcome.

DETAILED DESCRIPTION:
Patients with cutaneous tumors undergoing excision of either a biopsy-proven or a suspected cutaneous malignancy in the head and neck area were between April 2010 and November 2011 included in the trial. Patients were not included if they were less than 18 years old or if skin flaps or grafts were used. For patients with several cutaneous changes removed at the same time each excision was registered separately. The excisions were performed by 11 surgeons. Four surgeons performed 66% of all the procedures.

The assisting nurse documented data in a standardized form at wound closure. Patient factors such as age, sex, diabetes and corticoid treatment was recorded. The width and the length of the skin excision were measured, the number of sutures placed in the wound was counted and the size of the needle was documented. Whether wound edges were undermined or not, whether the excision was oriented in the natural skin tension line and whether subcuticular sutures were used or not was recorded. Skin closure was with monofilament nylon (Ehilon®) sutures (size 5.0 or 6.0). After the sutures were placed, adhesive tapes were placed perpendicular to the wound edges. The location of each wound was marked on a cartoon for later use at follow up. Patients were randomized in blocks of 8 to removal of sutures after either 7 or 14 days. Randomization was by opening sealed envelopes after wound closure.Thus the surgeons were blinded to the suture removal time.

All Participants received written information about wound care on which they were instructed not to wet the wound for 48 hour after the operation. After that they could take showers but not take baths until the sutures were removed. After suture removal new adhesive tapes were placed in the same manner as before and participants were informed to leave these in place for at least 7 days and also to protect the scar from sunlight for at least 6 months. For practical reasons patients with several excisions were randomized to one suture removal time. Sutures were removed at the surgical department conducting the trial.

Photographs were taken at one and twelve months after skin closure. Photographs of the wounds were taken in a standardized fashion at one month follow up by using a Canon EOS 550 by a research assistent. At the twelve month follow up the scar width was measured at three points in the scar and a mean value was calculated. The photographs at the twelve month follow up were taken by a professional photographer using Canon EOS Mark 2.

The images were assessed by two blinded otorhinolaryngologist an one blinded plastic surgeon all three stationed at University Hospitals. Each image was rated twice. A validated visual analogue scale (VAS) for overall cosmesis was used. The VAS is a 100-mm line with 0 representing the worst cosmetic outcome possible and 100 representing the best possible result. The minimum clinically important difference (MCID) of the 100-mm VAS is 10-25 mm. Using the line as a continuous entity, the surgeons marked the line, where it in their opinion best reflected the overall cosmetic outcome. The score was then measured in millimeters from the 0 point. Raters were instructed to take into account variables such as scar width, contour irregularities, step-off borders and presence of inflammation. Raters were also asked to note (twice) whether they noticed puncture marks in the scars or not.

This study had a power of 90% to discriminate with a MCID of 15-mm on the VAS for which 37 patients/scars were required in each group (p=0.05). This was based on using a standard deviation of 19.4 in a previous study using the VAS. Statistical analysis was performed with computer software (Microsoft Excel 2011 and SPSS) together with a statistician from the Department of Research and Development at Sundsvall hospital.

Ethical committee approval was granted for the study, and informed written consent was obtained before patient participation. The study was conducted at an Otorhinolaryngology division of the Surgical Center at Sundsvall Hospital receiving referrals from the dermatology division, primary health sector and private practicing otorhinolaryngologists (ORLs).

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing simple surgical excisions of suspected cutaneous malignancies in the head and neck and at least 18 years of age.

Exclusion Criteria:

* The use of local flaps or grafts.
* Not being able to understand the study protocol and the instructions given.
* Reoperation of the included wound/scar before study completion

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2011-04; Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Cosmetic assessment of scar | One month and one year
  assessment of scar with Visual Analog Cosmesis Scale after one month and one year. 3 blinded assessors.

SECONDARY OUTCOMES:
width of scar | one year
  with a mm-scale measure the width of the scar in 3 locations.

OTHER OUTCOMES:
Suture/puncture marks | One year

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Maleki, MD, Principal Investigator — Sundsvall Hospital; Eva Westman, MD, PhD, Study Director — Sundsvall Hospital, Umeå University
Locations (1):
- Sundsvall-Härnösand County Hospital, Sundsvall, Medelpad, Sweden